CLINICAL TRIAL: NCT02638272
Title: Outcomes of Radical Debridement Versus no Debridement Under Different Surgical Procedures for the Treatment of Thoracic and Lumbar Spinal Tuberculosis
Brief Title: Early Outcomes of Radical Debridement Versus no Debridement Under Different Surgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Qian Jun, Principal Investigator, The Second Hospital of Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1898
Record Dates: First submitted 2015-12-09; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Spinal Tuberculosis
MeSH Terms: conditions — Tuberculosis, Spinal

ARMS (1):
- spine surgery (Other): The objective was to compare the outcomes of radical debridement versus no debridement under different surgical procedures for the treatment of thoracic and lumbar tuberculosis.
  Interventions: Procedure: no debridement

INTERVENTIONS:
Procedure: no debridement — It is a spinal surgery performed with isolated posterior instrumentation without debridement.

SUMMARY:
Whether radical debridement is necessary for the treatment of thoracic and lumbar tuberculosis is still questionable. The objective of this prospective randomized study was to compare the outcomes of radical debridement versus no debridement under different surgical procedures for the treatment of thoracic and lumbar tuberculosis.

DETAILED DESCRIPTION:
Seventy-four thoracic and lumbar tuberculosis patients with a neurological function of grade D and E underwent surgeries from January 2009 to January 2014. All patients were divided into group A and group B by taking the drawing of lots. In group A, radical debridement, bone graft and instrumentation were performed. In group B, isolated posterior instrumentation without debridement were performed in all cases and drainage of iliopsoas abscess via laparoscopy in 2 cases. The operative time, blood loss, visual analogue score (VAS), erythrocyte sedimentation rate (ESR), kyphotic angle, Frankel grading, fusion rate and complications were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Frankel grading was grade D and E
2. Severe back pain
3. Abscess combined with high pressure symptoms
4. Larger sequestrum formation or sinus
5. Significant spinal instability.

Exclusion Criteria:

1. Frankel grading was grade A,B and C
2. Conservative treatment

Ages: 14 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2014-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The operative time in minutes | 5 years
blood loss in milliliter | 5 years
erythrocyte sedimentation rate (ESR) in mm/h | 5 years
kyphotic angle in degree | 5 years